CLINICAL TRIAL: NCT04508621
Title: A Phase 3, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of TNX-102 SL Taken Daily At Bedtime In Patients With Fibromyalgia
Brief Title: A Phase 3 Study To Evaluate The Efficacy And Safety Of TNX-102 SL In Patients With Fibromyalgia
Acronym: RALLY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-F306
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Fibromyalgia
Keywords: Pain; Sleep; Fibromyalgia; FM
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-102 SL Tablet, 5.6 mg (Experimental): 1 x TNX-102 SL 2.8 mg Tablet taken sublingually each day at bedtime for 2 weeks then 2 x TNX-102 SL 2.8 mg (5.6 mg) Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: TNX-102 SL
- Placebo SL Tablet (Placebo Comparator): 1 x Placebo Tablet taken sublingually each day at bedtime for 2 weeks then 2 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: Placebo SL Tablet

INTERVENTIONS:
Drug: TNX-102 SL — Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patient will have the dose increased to 2 tablets for 12 weeks.
  Other Names: Low dose cyclobenzaprine sublingual tablets
  Arms: TNX-102 SL Tablet, 5.6 mg
Drug: Placebo SL Tablet — Patients will take 1 tablet of randomly assigned study drug sublingually starting on Day 1 for 2 weeks. At the Week 2 visit, all patient will have the dose increased to 2 tablets for 12 weeks.
  Other Names: Placebo sublingual tablets
  Arms: Placebo SL Tablet

SUMMARY:
This is a Phase 3, randomized, parallel-group, double-blind, placebo-controlled, 14-week study designed to evaluate the efficacy and safety of TNX-102 SL 5.6 mg (2 x 2.8 mg tablets) taken daily at bedtime for the treatment of fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female 18 to 65 years of age, inclusive.
* The patient has a diagnosis of primary FM as defined by the 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria (American College of Rheumatology Preliminary Diagnostic Criteria)
* The in clinic 7-day recall NRS average daily pain intensity score at Screening Visit within protocol defined range.

Exclusion Criteria:

- History of or evidence for a diagnosis of borderline personality disorder (BPD).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, MD, Study Director — Tonix Pharmaceuticals, Inc.
Locations (36):
- United States (36):
  - Tonix Clinical Site, Birmingham, Alabama
  - Tonix Clinical Site, Phoenix, Arizona
  - Tonix Clinical Site, Oceanside, California
  - Tonix Clinical Site, San Diego, California
  - Tonix Clinical Site, Santa Ana, California
  - Tonix Clinical Site, Temecula, California
  - Tonix Clinical Site, Cromwell, Connecticut
  - Tonix Clinical Site, Fort Myers, Florida
  - Tonix Clinical Site, Jacksonville, Florida
  - Tonix Clinical Site, North Miami, Florida
  - Tonix Clinical Site, Ocala, Florida
  - Tonix Clinical Site, Orlando, Florida
  - Tonix Clinical Site, Alpharetta, Georgia
  - Tonix Clinical Site, Evansville, Indiana
  - Tonix Clinical Site, West Des Moines, Iowa
  - Tonix Clinical Site, Prairie Village, Kansas
  - Tonix Clinical Site, New Orleans, Louisiana
  - Tonix Clinical Site, Boston, Massachusetts
  - Tonix Clinical Site, Albuquerque, New Mexico
  - Tonix Clinical Site, Williamsville, New York
  - Tonix Clinical Site, High Point, North Carolina
  - Tonix Clinical Site, Raleigh, North Carolina
  - Tonix Clinical Site, Cincinnati, Ohio
  - Tonix Clinical Site, Dayton, Ohio
  - Tonix Clinical Site, North Canton, Ohio
  - Tonix Clinical Site, Oklahoma City, Oklahoma
  - Tonix Clinical Site, Tulsa, Oklahoma
  - Tonix Clinical Site, Portland, Oregon
  - Tonix Clinical Site, Warwick, Rhode Island
  - Tonix Clinical Site, Chattanooga, Tennessee
  - Tonix Clinical Site, Memphis, Tennessee
  - Tonix Clinical Site, Austin, Texas
  - Tonix Clinical Site, Dallas, Texas
  - Tonix Clinical Site, Salt Lake City, Utah
  - Tonix Clinical Site, Charlottesville, Virginia
  - Tonix Clinical Site, Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Started | 256 | 258
Completed | 189 | 210
Not Completed | 67 | 48
Not completed — Adverse Event | 39 | 16
Not completed — Lack of Efficacy | 2 | 8
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 10 | 14
Not completed — Lost to Follow-up | 12 | 9
Not completed — COVID-19 related crisis | 3 | 0
Not completed — Subject non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet | Total
Number analyzed (Participants) | 256 | 258 | 514
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (10.55) | 48.5 (10.60) | 48.7 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 245 | 487
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 16 | 24 | 40
  White | 226 | 223 | 449
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 256 | 258 | 514

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 14 in the Numerical Rating Scale (NRS) Weekly Average of Daily Self-reported Average Pain Severity Scores.
Description: Patients provide a daily numeric assessment of their average pain (24-hour recall), via an electronic diary, using an 11-point NRS. Scores range from 0 (no pain) to 10 (worst possible pain).
Time Frame: 14 weeks
Population: Intent to treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 256 | 258
score on a scale | -1.6 [-1.8 to -1.3] | -1.3 [-1.5 to -1.1]
Statistical Analysis 1: Comparison: TNX-102 SL Tablet, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.115, Mixed Model Repeated Measures; Multiple imputation used for missing data; LS Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.16 — Treatment difference = TNX-102 SL - Placebo

2. Secondary Outcome: Number of Patients With a Patient's Global Impression of Change (PGIC) Rating of "Very Much Improved" or "Much Improved"
Description: The PGIC is a fibromyalgia specific validated instrument on a scale of 1 to 7, where a score of 1 indicates the highest level of improvement and a score of 7 indicates a much worse outcome.
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Patients with missing data as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 256 | 258
Participants | 76 | 56
Statistical Analysis 1: Comparison: TNX-102 SL Tablet, 5.6 mg vs Placebo SL Tablet; Test type: Superiority — Patients with missing data considered non-responders; p = 0.038, Pearson Chi-Squared; Difference in Proportions = 8.0, 95% CI 2-sided [0.5 to 15.5]

3. Secondary Outcome: Change From Baseline to Week 14 in the Fibromyalgia Impact Questionnaire - Revised (FIQ-R) Symptoms Domain Score.
Description: The FIQ-R is a validated questionnaire. Scores on the symptoms domain range from 0 to 100 where a higher score means worse outcome.
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 256 | 258
score on a scale | -15.3 [-17.6 to -13.1] | -12.0 [-14.2 to -9.8]
Statistical Analysis 1: Comparison: TNX-102 SL Tablet, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.030, Mixed Model Repeated Measures; Multiple imputation used for missing data; LS Mean Difference = -3.4, 95% CI 2-sided [-6.4 to -0.3], Standard Error of Mean 1.55 — Treatment difference = TNX-102 SL - Placebo

4. Secondary Outcome: Change From Baseline to Week 14 in the FIQ-R Function Domain Score
Description: The FIQ-R is a validated questionnaire. Score on the function domain range from 0 to 90 where a higher score means worse outcome.
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 256 | 258
score on a scale | -8.8 [-10.9 to -6.7] | -8.4 [-10.5 to -6.4]
Statistical Analysis 1: Comparison: TNX-102 SL Tablet, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.797, Mixed Model Repeated Measures; Multiple imputation used for missing data; LS Mean Difference = -0.4, 95% CI 2-sided [-3.2 to 2.5], Standard Error of Mean 1.46 — Treatment Difference = TNX-102 SL - Placebo

5. Secondary Outcome: Change From Baseline to Week 14 in the Patient Reported Outcomes Measurement Information System (PROMIS) Score for Sleep Disturbance
Description: The PROMIS Sleep disturbance short form 8a consists of 8 questions on a 5-point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40.
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 256 | 258
score on a scale | -7.4 [-8.6 to -6.2] | -5.1 [-6.2 to -4.0]
Statistical Analysis 1: Comparison: TNX-102 SL Tablet, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.004, Mixed Model Repeated Measures; Multiple imputation used for missing data; LS Mean Difference = -2.3, 95% CI 2-sided [-3.8 to -0.7], Standard Error of Mean 0.80 — Treatment Difference = TNX-102 SL - Placebo

6. Secondary Outcome: Change From Baseline to Week 14 in the PROMIS Score for Fatigue
Description: The PROMIS fatigue short form 8a consist of 8 questions on a 5-point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40.
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 256 | 258
score on a scale | -6.6 [-7.7 to -5.5] | -5.4 [-6.4 to -4.3]
Statistical Analysis 1: Comparison: TNX-102 SL Tablet, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.101, Mixed Model Repeated Measures; Multiple imputation used for missing data; LS Mean Difference = -1.2, 95% CI 2-sided [-2.7 to 0.2], Standard Error of Mean 0.74 — Treatment Difference = TNX-102 SL - Placebo

7. Secondary Outcome: Change From Baseline to Week 14 in the Weekly Average of the Daily Diary Assessment of Sleep Quality
Description: Patients provide a daily numeric assessment of their sleep quality for the previous night, via an electronic diary, using an 11-point NRS. Scores range from 0 (best possible sleep) to 10 (worst possible sleep).
Time Frame: 14 weeks
Population: Intent to Treat population (all patients who were randomized). Multiple imputation for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
Number analyzed (Participants) | 256 | 258
score on a scale | -1.5 [-1.7 to -1.3] | -1.3 [-1.5 to -1.0]
Statistical Analysis 1: Comparison: TNX-102 SL Tablet, 5.6 mg vs Placebo SL Tablet; Test type: Superiority; p = 0.094, Mixed Model Repeated Measures; Multiple imputation used for missing data; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.16 — Treatment Difference = TNX-102 SL - Placebo

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | TNX-102 SL Tablet, 5.6 mg | Placebo SL Tablet
All-Cause Mortality (participants affected / at risk) | 0/256 | 0/258
Serious Adverse Events (participants affected / at risk) | 6/256 | 0/258
Other Adverse Events (participants affected / at risk) | 80/256 | 5/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablet, 5.6 mg (N=256) | Placebo SL Tablet (N=258)
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Localized infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-102 SL Tablet, 5.6 mg (N=256) | Placebo SL Tablet (N=258)
Hypoaesthesia oral (Gastrointestinal disorders) | 72 | 2
Oral discomfort (Gastrointestinal disorders) | 23 | 2
Tongue discomfort (Gastrointestinal disorders) | 16 | 2
Product taste abnormal (Product Issues) | 26 | 2

LIMITATIONS AND CAVEATS:
Recruitment during COVID-19 pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all study investigators.

DOCUMENTS (2):
  • Study Protocol (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04508621/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT04508621/SAP_001.pdf